CLINICAL TRIAL: NCT03680222
Title: Effect of Reversed Tracking Method of Stimulating Cricothyroid Muscles on the Identification and Protection of EBSLN in Thyroid Surgery
Brief Title: Effect of Reversed Tracking Method for Identification of EBSLN in Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, clinical professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IONM diffusion for EBSLN
Record Dates: First submitted 2018-09-09; First posted 2018-09-21 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Thyroid Cancer; Recurrent Laryngeal Nerve Injuries
Keywords: external branches of superior laryngeal nerve; thyroidectomy; thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Recurrent Laryngeal Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Different methods of protection of external branches of superior laryngeal nerve
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard method (No Intervention): Standard method recommended by the guide
- Reversed Tracking Method (Experimental): Reversed Tracking Method
  Interventions: Procedure: Reversed Tracking Method

INTERVENTIONS:
Procedure: Reversed Tracking Method — Reversed Tracking Method
  Arms: Reversed Tracking Method

SUMMARY:
The feasibility and effectiveness of Reversed Tracking Method for the identification and protection of extralaryngeal nerve branches in thyroid surgery were analyzed. Evidence-based medical evidence was used to evaluate the importance of EBSLN recognition and protection in thyroid surgery.

DETAILED DESCRIPTION:
The incidence of thyroid cancer in the world is growing rapidly. The current incidence of thyroid cancer in China is about 4.2/100,000, ranking the fourth in the incidence of female malignant tumors. Surgical treatment is the first and most important treatment for thyroid cancer. According to the existing literature, the injury rate of EBSLN in thyroid surgery can be as high as 58%. The quality of sound changes caused by EBSLN injury affects the quality of life of patients after surgery, and even affects the work and career of patients. therefore, seeking better EBSLN protection The method has great social and economic benefits.

ELIGIBILITY:
Inclusion criteria：

1. thyroid papillary cancer patients
2. thyroid adenoma patients
3. tumor diameter less than 4cm
4. patients who require only unilateral thyroid surgery as required by the guidelines

Exclusion criteria:

1. The upper pole tumor invades the anterior dorsum and may accumulate the area of the superior laryngeal nerve;
2. Patients who have previously performed head and neck surgery;
3. Preoperative laryngoscopy and sound assessment abnormalities or previous vocal cord surgery history;
4. If there is a language or hearing impairment, the follow-up assessment cannot be completed;
5. The assessment failure of nerve function due to the technical deficiency of the IONM equipment

Elimination criteria:

1. Patients with recurrent laryngeal nerve palsy after surgery affect the evaluation of the laryngeal nerve.
2. The patient is asked to withdraw from the follow-up assessment midway.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
The identification rate of the external branch of the superior laryngeal nerve. | up to 6 months postoperatively
  The identification rate of the external branch of the superior laryngeal nerve.

SECONDARY OUTCOMES:
Friedman classification | up to 6 months postoperatively
  Anatomical variability of the external branch of the superior laryngeal nerve according to Friedman classification.
videostrobolaryngoscopy | up to 6 months postoperatively
  The voice assessment included pre- and postoperative videostrobolaryngoscopy and analysis of maximum phonation time (MPT), voice level (VL), fundamental frequency (Fo), and voice quality rating on GRBAS scale.
analysis of maximum phonation time (MPT) | up to 6 months postoperatively
  The voice assessment included pre- and postoperative videostrobolaryngoscopy and analysis of maximum phonation time (MPT), voice level (VL), fundamental frequency (Fo), and voice quality rating on GRBAS scale.
voice level (VL) | up to 6 months postoperatively
  The voice assessment included pre- and postoperative videostrobolaryngoscopy and analysis of maximum phonation time (MPT), voice level (VL), fundamental frequency (Fo), and voice quality rating on GRBAS scale.
fundamental frequency (Fo) | up to 6 months postoperatively
  The voice assessment included pre- and postoperative videostrobolaryngoscopy and analysis of maximum phonation time (MPT), voice level (VL), fundamental frequency (Fo), and voice quality rating on GRBAS scale.
voice quality rating on GRBAS scale | up to 6 months postoperatively
  The voice assessment included pre- and postoperative videostrobolaryngoscopy and analysis of maximum phonation time (MPT), voice level (VL), fundamental frequency (Fo), and voice quality rating on GRBAS scale.

CONTACTS AND LOCATIONS:
Overall Officials: wenxin zhao, md, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No